CLINICAL TRIAL: NCT01068275
Title: Lumbar Plexus Catheter Versus Femoral Nerve Catheter Versus Single-shot Femoral Block for Postoperative Pain Control After Anterior Cruciate Ligament Reconstruction
Brief Title: Lumbar Plexus Catheter Versus Femoral Nerve Catheter for Postoperative Pain After Anterior Cruciate Ligament (ACL) Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Felicia Birch, M.D., Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCHAnes1
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2010-08-26 (Estimated); Status verified 2010-08

CONDITIONS: Postoperative Pain
Keywords: anterior cruciate ligament; pain, postoperative; peripheral nerve catheter; nerve block; Children undergoing anterior cruciate ligament repair
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lumbar plexus catheter (Active Comparator)
  Interventions: Procedure: lumbar plexus catheter
- femoral nerve catheter (Active Comparator)
  Interventions: Procedure: femoral nerve catheter
- single-shot femoral block (Active Comparator)
  Interventions: Procedure: single-shot femoral block

INTERVENTIONS:
Procedure: lumbar plexus catheter — lumbar plexus catheter with 0.2% ropivacaine at 0.15 ml/kg/hr (max 10 ml/hr)
  Other Names: psoas compartment catheter
  Arms: Lumbar plexus catheter
Procedure: femoral nerve catheter — femoral nerve catheter with 0.2% ropivacaine at 0.15 ml/kg/hr (max 10 ml/hr)
  Arms: femoral nerve catheter
Procedure: single-shot femoral block — single-shot femoral block with 0.2% ropivacaine 0.3 ml/kg (max 20 ml)
  Arms: single-shot femoral block

SUMMARY:
Randomized trial comparing lumbar plexus catheter versus femoral nerve catheter (single-shot femoral block as control group) for postoperative pain control after anterior cruciate ligament repair in children (age 11-21). Primary outcome is pain scores for the first 72 hours. Secondary outcomes include opioid consumption, incidence of opioid side effects and quality of recovery (previously validated scale). Our hypothesis is that lumbar plexus catheter will provide superior pain control and overall quality of recovery compared to femoral nerve catheters.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-2
* Age 11-21
* Undergoing anterior cruciate ligament repair

Exclusion Criteria:

* Patient refusal
* Coagulopathy
* Systemic infection or infection at needle insertion site
* Allergy to ropivacaine or opioids
* Taking chronic opioids
* Unavailable by phone

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 114 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain scores | 72 hours

SECONDARY OUTCOMES:
Quality of recovery | 72 hours
Opioid consumption | 72 hours
Opioid side effects | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Felicia M Birch, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States